CLINICAL TRIAL: NCT04186819
Title: A Prospective, Phase 3, Multi Center, Single-arm, Imaging Study Investigating the Safety and Diagnostic Performance of rhPSMA 7.3 (18F) Positron Emission Tomography (PET) Ligand in Men With Newly Diagnosed Prostate Cancer
Brief Title: Imaging Study to Investigate the Safety and Diagnostic Performance of rhPSMA 7.3 (18F) in Newly Diagnosed Prostate Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Blue Earth Diagnostics (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BED-PSMA-301
Record Dates: First submitted 2019-11-22; First posted 2019-12-05 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: Primary Prostate Cancer; Diagnostic; Prostate Specific Membrane Antigen (PSMA); Positron Emission Tomography (PET) Scan
MeSH Terms: conditions — Prostatic Neoplasms; Disease | interventions — Injections; Positron-Emission Tomography

STUDY DESIGN:
Intervention Model Description: Positron Emission Tomography (PET) Imaging study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Single intravenous administration of rhPSMA-7.3 (18F) for PET Scan
  Interventions: Drug: rhPSMA-7.3 (18F) Injection; Diagnostic Test: Positron Emission Tomography scan

INTERVENTIONS:
Drug: rhPSMA-7.3 (18F) Injection — Radioligand for PET CT scanning
  Other Names: No other interventions
Diagnostic Test: Positron Emission Tomography scan — imaging test with radioligand
  Other Names: PET scan

SUMMARY:
A prospective, Phase 3, multi center, single-arm, imaging study investigating the safety and diagnostic performance of Radio-hybrid Prostate Specific Membrane Antigen (rhPSMA) 7.3 (18F) Positron Emission Tomography (PET) ligand in men with newly diagnosed prostate cancer.

DETAILED DESCRIPTION:
Main objective is to assess the sensitivity and specificity of rhPSMA-7.3 (18F) positron emission tomography (PET) in detecting N1 disease (as determined by the central blinded image evaluation [BIE]) on a patient level compared to the histopathology of pelvic lymphatic tissue removed during radical prostatectomy (RP) and pelvic lymph node dissection (PLND). At least one positive pelvic LN on PET (N1) and one positive lymph node (LN) as determined by histopathology (pN1) on the same side of the pelvis (left or right) will be deemed a True Positive (TP) at the patient level.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male and aged >18 years old.
2. Histologically confirmed adenocarcinoma of the prostate.
3. Patients electing to undergo Radical Prostatectomy (RP) with Pelvic lymph node dissection (PLND).

Exclusion Criteria:

1. Patients who are planned to have an x-ray contrast agent or other PET radiotracer <24 hours prior to the PET scan.
2. Patients currently receiving, or with a prior history of, Androgen Deprivation Therapy (ADT).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients required to have unfavorable intermediate-, high-risk or very high-risk Prostate Cancer
Enrollment: 356 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (29):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Tower Urology, Los Angeles, California
  - University of California Irvine Medical Center (UCIMC), Orange, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Emory University Hospital, Atlanta, Georgia
  - Northside Hospital, Austell, Georgia
  - NorthShore University HealthSystem, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Richard L Roudebush VA Medical Center, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - The Urologic Institute of Northeastern New York - Community, Albany, New York
  - Queens Hospital Center (QHC) - Queens Cancer Center, Jamaica, New York
  - Mount Sinai Faculty Practice Associates, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Montefiore Hospital, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - MidLantic Urology, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - MD Anderson Hospital, Houston, Texas
  - Urology San Antonio, San Antonio, Texas
  - University of Virginia - Health Science Center, Charlottesville, Virginia
  - Virginia Oncology Associates PC, Norfolk, Virginia
- Turku University Hospital, Turku, Finland
- Germany (2):
  - Klinik und Poliklinik fur Urologie, Hamburg
  - TU München, Munich
- Netherlands (2):
  - CWZ, Nijmegen
  - Maxima MC, Veldhoven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Surasi DS, Eiber M, Maurer T, Preston MA, Helfand BT, Josephson D, Tewari AK, Somford DM, Rais-Bahrami S, Koontz BF, Bostrom PJ, Chau A, Davis P, Schuster DM, Chapin BF; LIGHTHOUSE Study Group. Diagnostic Performance and Safety of Positron Emission Tomography with 18F-rhPSMA-7.3 in Patients with Newly Diagnosed Unfavourable Intermediate- to Very-high-risk Prostate Cancer: Results from a Phase 3, Prospective, Multicentre Study (LIGHTHOUSE). Eur Urol. 2023 Oct;84(4):361-370. doi: 10.1016/j.eururo.2023.06.018. Epub 2023 Jul 5. PMID 37414702

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was from 02 Mar 20 (first patient, screening visit) and 18 Feb 22 (database lock), with the last patient, last visit on 21 Jun 21. It was conducted at 34 activated study sites (31 recruited) in 4 countries. Of the 372 patients screened, 356 patients met all the study eligibility criteria. 16 patients were screen failures so not included
Pre-assignment Details: Baseline safety evaluations performed at screening (Visit 1) comprised vital signs, focused physical examination and recording of any adverse events (AEs) from the time of informed consent.
Period: Overall Study
Arm/Group | Patients
Started | 356
Completed | 336
Not Completed | 20
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Opted for EBRT | 1
Not completed — Opted SBRT | 1
Not completed — Patient decided to have focal ablation and not surgery | 2
Not completed — Physician Decision | 1
Not completed — RP Delayed | 1
Not completed — Sponsor Decision: Outdated FU Timeline | 1
Not completed — Subject declined for financial reasons | 1
Not completed — The subject declined any biopsy or surgery due to COVID-19 pandemic | 1
Not completed — The subject declined for any biopsy or other imaging | 2
Not completed — The subject opted for other treatment option | 2
Not completed — The subject opted for other treatment options | 1
Not completed — Withdrawal by Subject | 3
Not completed — Reason not specified | 1

BASELINE CHARACTERISTICS:
Population: The FAS comprised 356 patients who were scheduled to receive the rhPSMA-7.3 (18F) injection and met the inclusion/exclusion criteria
Groups:
- Single Arm: Single intravenous administration of rhPSMA-7.3 (18F) for PET Scan
  rhPSMA-7.3 (18F) Injection: Radioligand for PET CT scanning
  Positron Emission Tomography scan: imaging test with radioligand
Arm/Group | Single Arm
Number analyzed (Participants) | 356
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (6.98)
Age, Customized [Number; unit: participants] — Age in years split into 2 groups
  participants
    < 65 years | 163
    ≥ 65 years | 193
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 356
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity split into 2 substantive groups and those for whom it was not reported
  Participants
    Hispanic or Latino | 17
    Not Hispanic or Latino | 311
    Unknown or Not Reported | 28
Race/Ethnicity, Customized [Number; unit: participants] — Race split into 3 substantive categories and also those for whom it was not reported
  participants
    Black or African American | 30
    White | 289
    Other | 4
    Not Reported | 33
Region of Enrollment [Number; unit: participants]
  Netherlands | 14
  United States | 238
  Finland | 18
  Germany | 86
Total Gleason Score [Number; unit: participants] — Gleason score (defined by the International Society of Urological Pathologists) was based on prostate biopsy.
  Score 6 - The cells look similar to normal prostate cells. The cancer is likely to grow very slowly, if at all
  Score 7 - Most cells still look similar to normal prostate cells. The cancer is likely to grow slowly
  Score 8 - Some cells look abnormal. The cancer might grow quickly or at a moderate rate
  Score 9 or 10 - The cells look very abnormal. The cancer is likely to grow quickly
  participants
    =7 | 160
    =8 | 87
    =9 | 97
    =10 | 6
    ≤ 6 | 6
TNM (Tumor-Node-Metastasis) Stage T [Number; unit: participants] — Tumour (T) describes the size or area of the cancer
  T1 means the cancer is too small to be seen on a scan, or felt during an examination of the prostate
  T1a means that the cancer is in less than 5% of the removed tissue
  T1c cancers are found by biopsy, for example after a raised PSA level
  T2 means the cancer is completely inside the prostate gland
  T3a means the cancer has broken through the capsule (covering) of the prostate gland
  T3b means the cancer has spread into the tubes that carry semen (seminal vesicles)
  T4 means the cancer has spread into other body organs nearby
  participants
    T1 | 16
    T1a | 2
    T1c | 127
    T2 | 58
    T2a | 18
    T2b | 25
    T2c | 33
    T3 | 20
    T3a | 21
    T3b | 12
    T3c | 1
    T4 | 2
    TX | 9
    Missing | 12
Gleason Grade Group (GGG) [Number; unit: participants] — GGG (defined by the International Society of Urological Pathologists) was based on prostate biopsy.
  Group 1: The cells look similar to normal prostate cells. The cancer is likely to grow very slowly, if at all
  Group 2: Most cells still look similar to normal prostate cells. The cancer is likely to grow slowly
  Group 3: The cells look less like normal prostate cells. The cancer is likely to grow at a moderate rate
  Group 4: Some cells look abnormal. The cancer might grow quickly or at a moderate rate
  Group 5: The cells look very abnormal. The cancer is likely to grow quickly
  participants
    =1 | 6
    =2 | 50
    =3 | 110
    =4 | 87
    =5 | 103
TNM Stage M [Number; unit: participants] — Metastasis (M) describes whether the cancer has spread to a different part of the body.
  M0 means the cancer hasn't spread to other parts of your body.
  M1 means the cancer has spread to other parts of the body outside the pelvis. It is split into M1a, M1b and M1c.
  M1a means there are cancer cells in lymph nodes outside the pelvis
  M1b means there are cancer cells in the bone
  M1c means there are cancer cells in other parts of the body such as the lungs
  participants
    M0 | 290
    M1 | 4
    M1a | 1
    M1b | 1
    MX | 48
    Missing | 12
Prostate-specific antigen (PSA) Characterization (ng/mL) [Number; unit: participants]
  >1.0 to 2.0 | 2
  >2.0 to 5.0 | 62
  >5.0 to 10.0 | 134
  >10.0 | 158
Baseline Risk Category [Number; unit: participants] — Baseline Risk Category. High-risk or Very-high risk defined as meeting any one of these criteria: T-stage T3 (including T3a and T3b) or T4, GGG 4 or 5, Primary Gleason pattern 5, or PSA >20 ng/mL.
  participants
    High-risk or Veryhigh-risk | 241
    Immediate-Risk | 115
TNM Stage N [Number; unit: participants] — Node (N) describes whether the cancer has spread to the lymph nodes.
  N0 means that the nearby lymph nodes don't contain cancer cells
  N1 means there are cancer cells in lymph nodes near the prostate
  participants
    N0 | 284
    N1 | 11
    NX | 49
    Missing | 12
Body Mass Index [Mean (Standard Deviation); unit: Kg/m2] — Body mass index on Day 1 (Kg/m2) Population: Number analyzed differs from overall due to missing data.
  Kg/m2
    number analyzed (Participants) | 334
    (all) | 28.20 (4.341)
Time since initial cancer diagnosis [Mean (Standard Deviation); unit: months] — Time since initial cancer diagnosis relative to the date of informed consent.
  months | 2.9 (10.27)
Time since last PSA Measurement [Mean (Standard Deviation); unit: months] — Population: Number analyzed differs from overall due to missing data.
  months
    number analyzed (Participants) | 354
    (all) | 2.5 (2.83)
Last PSA Measurement (ng/mL) [Mean (Standard Deviation); unit: ng/mL] | 15.090 (18.2450)

OUTCOME MEASURES:

1. Primary Outcome: Specificity
Description: The primary objective of the study is to assess the sensitivity and specificity of rhPSMA-7.3 (18F) positron emission tomography (PET) in detecting N1 disease (as determined by the central BIE) on a patient level compared to the histopathology of pelvic lymphatic tissue removed during RP and PLND.
Time Frame: Conventional images within 60 days or at least 24 hours prior to rhPSMA-7.3 (18F) PET, followed by treatment within 60 days post IMP administration
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Efficacy Analysis Population: All patients who received rhPSMA-7.3 (18F) injection followed by a PET/CT scan and who underwent RP and PLND
Arm/Group | Efficacy Analysis Population
Number analyzed (Participants) | 226
percentage
  Central Reader 1 | 92.9 [88.8 to 95.9]
  Central Reader 2 | 93.8 [89.8 to 96.6]
  Central Reader 3 | 96.9 [93.7 to 98.7]

2. Primary Outcome: Sensitivity
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Efficacy Analysis Population
Number analyzed (Participants) | 70
percentage
  Central Reader 1 | 30 [19.6 to 42.1]
  Central Reader 2 | 27.1 [17.2 to 39.1]
  Central Reader 3 | 22.9 [13.7 to 34.4]

3. Secondary Outcome: Verified Detection Rate (VDR) for M1 Lesions - Percentage of Patients in Whom rhPSMA-7.3 (18F) Imaging Detected at Least One Verified M1 Metastasis, as Determined by Central BIE and Confirmed by SoT (Biopsy or Imaging) (Objective 1)
Description: This was a key secondary endpoint in this study and included patients in the EEP with rhPSMA-7.3 (18F) imaging.
Time Frame: Conventional images within 60 days or at least 24 hours prior to rhPSMA-7.3 (18F) PET. followed by treatment within 60 days post IMP administration
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Extended Efficacy Population (EEP): all patients who received rhPSMA-7.3 (18F) injection followed by a PET scan. This population included M0 and M1 patients independent of performance of RP and PLND and was used for M1 related efficacy and Kappa statistics.
Arm/Group | Extended Efficacy Population (EEP)
Number analyzed (Participants) | 352
percentage
  Central Reader 1 | 9.9 [7.0 to 13.6]
  Central Reader 2 | 14.2 [10.7 to 18.3]
  Central Reader 3 | 10.2 [7.3 to 13.9]

4. Secondary Outcome: Percentage of Patients With Negative Conventional Imaging for M1 Disease in Whom rhPSMA-7.3 (18F) PET Detected at Least One Verified M1 Metastasis, as Determined by Central BIE (Objective 2)
Description: Patients counted in this variable were a subset of those in Point 1 above, where both the numerator and denominator were only counting patients with negative conventional imaging (according to investigator assessment) for M1 disease.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Extended Efficacy Population (EEP)
Number analyzed (Participants) | 331
percentage
  Central Reader 1 | 8.8 [5.9 to 12.3]
  Central Reader 2 | 13.0 [9.6 to 17.1]
  Central Reader 3 | 8.5 [5.7 to 12.0]

5. Secondary Outcome: Patient-level PPV of rhPSMA-7.3 (18F) PET BIE for N1 and M1 Lesions Compared to Histopathology or Confirmatory Imaging (M1 Lesions Only) (Objective 3)
Description: This analysis included patients with rhPSMA-7.3 (18F) imaging and either N1 or M1 lesions detected, where PPV=TP/(TP+FP).
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Efficacy Analysis Population (EAP): N1 lesions compared to histopathology
- Extended Efficacy Population (EEP): M1 lesions compared to histopathology or confirmatory imaging
Arm/Group | Efficacy Analysis Population (EAP) | Extended Efficacy Population (EEP)
Number analyzed (Participants) | 296 | 352
percentage
  Central Reader 1 | 56.8 [39.5 to 72.9] | 62.5 [48.5 to 75.1]
  Central Reader 2 | 57.6 [39.2 to 74.5] | 51.0 [40.7 to 61.3]
  Central Reader 3 | 69.6 [47.1 to 86.8] | 57.1 [44.0 to 69.5]

6. Secondary Outcome: PPV of rhPSMA-7.3 (18F) PET for Detecting PLN Metastases Compared to Surgical Pathology on a Patient-level, in Which a FP Patient is Defined as Having at Least One FP Region (Right or Left Pelvis), Regardless of Any Coexisting TP Findings (Objective 4)
Description: This analysis included patients in the EAP where rhPSMA-7.3 (18F) imaging detected PLN metastasis. Regions where rhPSMA7.3 (18F) imaging detected no LN metastasis were not included (by definition of PPV), hence only TP and FP regions were considered. TPs were all patients with a surgical pathology confirmed positive region and without a FP region. FP patients were those patients with any rhPSMA7.3 (18F) PETpositive region with negative or no surgical pathology.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Efficacy Analysis Population (EAP): All patients who received rhPSMA-7.3 (18F) injection followed by a PET/CT scan and who underwent RP and PLND
Arm/Group | Efficacy Analysis Population (EAP)
Number analyzed (Participants) | 296
percentage
  Central Reader 1 | 48.6 [31.9 to 65.6]
  Central Reader 2 | 54.5 [36.4 to 71.9]
  Central Reader 3 | 65.2 [42.7 to 83.6]

7. Secondary Outcome: NPV of rhPSMA-7.3 (18F) PET for Detecting PLN Metastases Compared to Surgical Pathology on a Patient-level, in Which a FN Patient is Defined as Having at Least One FN Region (Right or Left Pelvis), Regardless of Any Coexisting TN Findings (Objective 5)
Description: This analysis included patients in the EAP with rhPSMA-7.3 (18F) imaging where no LN metastases were detected and LN surgical pathology was available; where NPV=TN/(TN+FN).
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Efficacy Analysis Population (EAP)
Number analyzed (Participants) | 296
percentage
  Central Reader 1 | 81.3 [76.3 to 85.7]
  Central Reader 2 | 80.8 [75.8 to 85.2]
  Central Reader 3 | 79.9 [74.8 to 84.4]

8. Secondary Outcome: The Percentage of Patients Being Upstaged to N1 or M1 Disease. (Objective 6a)
Description: TP [confirmed by SoT] central BIE PET finding and negative conventional imaging finding from the local reading
Time Frame: as for outcome 1
Measure: Number; unit: percentage
Groups:
- Upstaged to N1: Percentage of patient being upstaged to N1 (EEP)
- Upstaged to M1: Percentage of patient being upstaged to M1 (EEP)
Arm/Group | Upstaged to N1 | Upstaged to M1
Number analyzed (Participants) | 352 | 352
percentage
  Central Reader 1 | 5.1 | 8.2
  Central Reader 2 | 4.3 | 12.2
  Central Reader 3 | 3.7 | 8.0

9. Secondary Outcome: The Percentage of Patients in Whom Planned RP Was Converted to EBRT. (Objective 6b)
Time Frame: as for outcome 1
Measure: Number; unit: percentage
Arm/Group | Extended Efficacy Population (EEP)
Number analyzed (Participants) | 352
percentage | 2.6

10. Secondary Outcome: Kappa Statistic for the Agreement Between and Within Blinded Independent Readers on the Interpretation of rhPSMA-7.3 (18F) Scans (Objective 7)
Description: Pairwise agreement between any 2 of the 3 readers (Kappa statistic could not be calculated for 2 of the pairwise agreements), and within readers between the initial read and re-read (Kappa statistics could not be calculated for 2 of the within-reader agreements)
Time Frame: PET/CT scans on Day 1
Population: All patients who received rhPSMA-7.3 (18F) injection followed by a PET/CT scan
Measure: Number; unit: percentage
Groups:
- Extended Efficacy Population (EEP): All patients who received rhPSMA-7.3 (18F) injection followed by a PET/CT scan
Arm/Group | Extended Efficacy Population (EEP)
Number analyzed (Participants) | 352
percentage
  Agreement between reader 1 and reader 2 | 97.7
  Agreement between Reader 1 and Reader 3 | 95.2
  Agreement between Reader 2 and Reader 3 | 96.9
  Agreement between initial read and re-read in Reader 1 | 100
  Agreement between initial read and re-read in Reader 2 | 100
  Agreement between initial read and re-read in Reader 3 | 95.7

ADVERSE EVENTS:
Time Frame: All AEs were recorded throughout the study from informed consent through study completion, an average of 60 days post-IMP administration.
Description: AEs were coded using MedDRA and data listed by patient, including study site, patient identifier, age, race, AE (MedDRA SOC, PT and verbatim term), dates of onset and resolution, duration, CTCAE toxicity grade, seriousness, action taken, outcome and causality. Deaths, SAEs and AEs leading to discontinuation were also listed by patient
Groups:
- Full Safety Population (FSP): All patients who received the rhPSMA-7.3 (18F) injection. The FSP was used for all safety summaries.
Arm/Group | Full Safety Population (FSP)
All-Cause Mortality (participants affected / at risk) | 0/356
Serious Adverse Events (participants affected / at risk) | 0/356
Other Adverse Events (participants affected / at risk) | 28/356
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Safety Population (FSP) (N=356)
Tracheal deviation (Injury, poisoning and procedural complications) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Thrombophlebitis (Vascular disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (5)
Chills (General disorders) | 1 (1)
Injection site pain (General disorders) | 3 (3)
Peripheral swelling (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Nervousness (Psychiatric disorders) | 1 (1)
Haematuria traumatic (Renal and urinary disorders) | 1 (1)
Lower urinary tract symptoms (Renal and urinary disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT04186819/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT04186819/SAP_002.pdf